CLINICAL TRIAL: NCT04733703
Title: Impact of Postanesthesia Care Unit Delirium on Postoperative Quality of Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PACQoR 2
Record Dates: First submitted 2020-09-28; First posted 2021-02-02 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Neurocognitive Disorders; Delirium; Postoperative Recovery; Anesthesia
MeSH Terms: conditions — Delirium | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — assessment of postoperative quality of recovery with the QoR-15

SUMMARY:
Postanesthesia care unit (PACU) delirium is subtype of postoperative delirium that occurs early after anesthesia and surgery during the recovery period. The consequences of PACU delirium have not been investigated thoroughly. So far it is unknown, whether patients with PACU delirium experience impaired postoperative quality of recovery.

The aim of this observational study is to assess the impact of PACU delirium on quality of recovery 24 hours after general anesthesia for elective non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* general anesthesia
* fluency in German

Exclusion Criteria:

* expected postoperative ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are scheduled for elective non-cardiac surgery and who will receive general anesthesia, are eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
postoperative quality of recovery | 24 hours postoperatively
  patient-reported quality of recovery after surgery and anesthesia with the QoR-15, ranging from 0 (poor recovery) to 150 (excellent recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fischer, MD, PhD, Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No